CLINICAL TRIAL: NCT04145310
Title: A Prospective, Single-Center, Double-Blind, Placebo-Controlled Trial of BOL-DP-o-04 in Patients With Low Back Pain and Sciatica
Brief Title: BOL-DP-o-04 in Patients With Low Back Pain and Sciatica
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Breath of Life International Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOL-P-11
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain; Sciatica
MeSH Terms: conditions — Low Back Pain; Sciatica

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: BOL-DP-o-04 + SCO
- Arm B (Placebo Comparator)
  Interventions: Drug: Placebo + SCO

INTERVENTIONS:
Drug: BOL-DP-o-04 + SCO — sublingual drops
  Arms: Arm A
Drug: Placebo + SCO — sublingual drops
  Arms: Arm B

SUMMARY:
The study is aimed to evaluate the pain-relieving effect of BOL-DP-o-04, in addition to SOC, on Low Back Pain and Sciatica.

DETAILED DESCRIPTION:
A Prospective, Single-Center, Double-Blind, Placebo-Controlled Trial of BOL-DP-o-04 in Patients with Low Back Pain and Sciatica. The study is aimed to evaluate the pain-relieving effect of BOL-DP-o-04, in addition to SOC, on Low Back Pain and Sciatica.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Mild to Severe Low Back Pain and/or Sciatica
3. Imaging studies (CT or MRI) supporting anatomical abnormality that could be the cause of the symptoms
4. Must be physically and mentally willing and able to comply with the treatment regimen and understand the informed consent and study procedures
5. Signed and dated Informed Consent Form (ICF)
6. Non-responsive to standard therapy for at least 1 month

Exclusion Criteria:

1. VAS Pain Subscale score at Screening is less than 6 (with 0 being no pain and 10 being worse imaginable pain)
2. Known allergy to cannabis or its components
3. A patient who is pregnant or intends to become pregnant during the study
4. A patient who is nursing or intends to nurse during the study
5. A patient suffering from a mental disorder precluding administration of study drug
6. Prisoners
7. A Patient is unable to sign an informed consent form
8. Unstable angina pectoris
9. Cardiac insufficiency precluding cannabis administration
10. Immunosuppressed patients unless BOL-DP-o-04 administration is deemed safe by the treating physician
11. Known Aspergillus infection
12. Panic attacks or anxiety unless a psychiatrist allowed BOL-DP-o-04 following intake interview
13. Any mental/psychiatric illness in first-degree relative in a young patient < 30-year-old.
14. Patient with congestive heart failure
15. Subjects who get the following medications: opiates, Primidone, Phenobarbitol, arbamazepine, Rifampicin, Rifabutin, Troglitazone, and Hypericum perforatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline to Day 114
  Change in the Oswestry Disability Index. The questionnaire is composed by 10 sections Each section can be scored 0 to 5, 5 being the worst case. The score is calculated by summing the different sections and then doubling the total. Maximum score is 100.

SECONDARY OUTCOMES:
Brief Pain Index | Baseline to Day 100
  Change in the Brief Pain Index relative to baseline. The Brief Pain Inventory rapidly assesses the severity of pain and its impact on functioning
Short Form (SF12) Mental | Screening to Day 100
  Change in Short Form (SF12) Mental Composite Score.The SF-12 consists of a subset of 12 items that measure eight health domains to assess physical and mental health
Pittsburgh Sleep Quality Index | Screening to Day 100
  Change in Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score
Opiate consumption and analgesic medication consumption | Screening to Day 100
  Change in Opiate consumption and analgesic medication consumption
Patient Global Impression | Baseline to Day 100
  Change in Patient global impression. The Patient Global Impression is a 7 point scale depicting a patient's rating of overall improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No